CLINICAL TRIAL: NCT03149172
Title: Comparison of Post Tooth Extraction Healing Using Different Xenograft Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Yong Hur, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #10963
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The surgeon and the subject will not be blinded. The evaluation of the core histology will be done by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Equimatrix® (Experimental): Equimatrix® + Mucograft or alternatives
  Interventions: Device: Equimatrix®
- Bio-Oss® (Experimental): Bio-Oss® + Mucograft or alternatives
  Interventions: Device: Bio-Oss®
- Endobon® (Experimental): Endobon® + Mucograft or alternatives
  Interventions: Device: Endobon®

INTERVENTIONS:
Device: Equimatrix® — Ridge preservation bone grafting after tooth extraction
  Arms: Equimatrix®
Device: Bio-Oss® — Ridge preservation bone grafting after tooth extraction
  Arms: Bio-Oss®
Device: Endobon® — Ridge preservation bone grafting after tooth extraction
  Arms: Endobon®

SUMMARY:
The purpose of this pilot study is to conduct a interventional prospective clinical trial to evaluate the efficacy of three different xenografts for ridge preservation by comparing the quality of newly formed bone using histomorphometric and micro CT analysis.The three xenograft materials under investigation are Bio-Oss® (bovine derived xenograft), Equimatrix® (equine derived xenograft), and Endobon® (bovine derived xenograft). There are no prospective studies comparing the effectiveness of these three materials, Bio-Oss®, Endobon® and Equimatrix®, when placed in extraction sockets.

Participants will be recruited from patients in the TUSDM clinics that require extraction of single rooted non-molar tooth and are treatment planned to receive dental implants in the future. Participants will be randomized to receive one of the three xenograft materials after tooth extraction. The percentage of newly formed bone and bone density will be compared between the three materials 4-6 months after ridge preservation.

DETAILED DESCRIPTION:
This is a pilot prospective clinical trial in which histological and micro CT analysis will be utilized to compare between Endobon®, Equimatrix®, and Bio-Oss®.

Primary aim: Compare the percentage of newly formed bone between Equimatrix®, Bio-Oss® and Endobon®.

The investigators hypothesize that the mean percentage of newly formed bone from Equimatrix® will be higher than Bio-Oss® and/or Endobon®.

Secondary aim: Compare the bone density between Equimatrix®, Bio-Oss® and Endobon®.

The investigators hypothesize that the bone density from Equimatrix® will be higher than Bio-Oss® and/or Endobon®.

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable single rooted tooth in anterior or premolar region
* Patient previously treatment planned for implant procedure and implant restoration.
* > 10 mm from maxillary sinus or inferior alveolar canal (IAC)
* Intact buccal bone (only minor dehiscence or fenestrations (approximately < 50% of socket depth) can be accepted
* Non-smokers.
* Patients treatment planned for extraction and ridge preservation at Tufts University School of Dental Medicine.

Exclusion Criteria:

* Poor oral hygiene (plaque index>30%).
* Systemic diseases that affect bone metabolism:

  i. Osteoporosis ii. Osteomalacia iii. Hyperthyroidism iv. Hyperparathyroidism v. Paget's disease
* Inflammatory and autoimmune diseases of the oral cavity (severe bone loss) (self-report):

  i. Severe chronic periodontitis ii. Aggressive periodontitis iii. Necrotizing ulcerative periodontitis iv. Crohn's disease v. Multiple sclerosis vi. Rheumatoid arthritis vii. Systemic lupus erythematosus
* History of radiation to the head and neck, and /or chemotherapy.
* Current corticosteroid therapy.
* History of IV Bisphosphonates therapy or >3 years of oral intake.
* Infectious diseases such as HIV, tuberculosis, Hepatitis (self-report).
* Known allergy to research related materials.
* Self-reported pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Hur, DDS, DMD, MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 subjects were screened. However, only 21 subjects were enrolled. 4 patients didn't participate the study.
Period: Overall Study
Arm/Group | Equimatrix® | Bio-Oss® | Endobon®
Started | 8 | 6 | 7
Completed | 6 | 5 | 5
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Equimatrix® | Bio-Oss® | Endobon® | Total
Number analyzed (Participants) | 8 | 6 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 7 | 16
  >=65 years | 3 | 2 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.7) | 55.2 (12.6) | 53.5 (7.1) | 56.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 5 | 3 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percent New Bone Formation
Description: Histomorphometric determination of % new bone formation
Time Frame: 4-6 months after ridge preservation surgery
Measure: Mean (Standard Deviation); unit: percentage of new bone formation
Arm/Group | Equimatrix® | Bio-Oss® | Endobon®
Number analyzed (Participants) | 6 | 5 | 5
percentage of new bone formation | 41 (30) | 25 (18) | 26 (26)

2. Secondary Outcome: Bone Density
Description: Measured by Micro CT Scanning
Time Frame: 4-6 months after ridge preservation surgery
Population: The micro-CT data was anaylzed as a preliminary outcome of the primary outcome. A total of 10 patient data was used.
Measure: Mean (Standard Deviation); unit: percentage of bone volume
Arm/Group | Equimatrix® | Bio-Oss® | Endobon®
Number analyzed (Participants) | 3 | 3 | 4
percentage of bone volume | 25.6 (18.7) | 23.0 (7.9) | 12.9 (11.1)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were recorded in source documents and on case report forms. All adverse events were recorded, monitored, and reported to the IRB at time of continuing review or at the study's termination. None of the participants had adverse events to report during the study period.
Arm/Group | Equimatrix® | Bio-Oss® | Endobon®
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No